CLINICAL TRIAL: NCT03330158
Title: Clinical Assessment of a Motorized Spinal Distraction Rod in the Severe to Early Scoliosis Child
Acronym: ASTS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC31/15/7851
Record Dates: First submitted 2016-07-11; First posted 2017-11-06 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ASTS device (Experimental): Implantation of device ASTS (for ACTIVE TREATMENT SCOLIOSIS SYSTEM ) in children between 4 and 10
  Interventions: Device: ASTS

INTERVENTIONS:
Device: ASTS — Implantation of a motorized spinal distraction rod

SUMMARY:
The purpose of this biomedical research is to evaluate the feasibility of the treatment with the new spinal distraction device ASTS in patients aged 4 to 10 years with severe early onset scoliosis.

The hypothesis of this project is that the new fully implantable motorized spinal distraction device may provide a correction of scoliosis and progressive elongation ensuring patient comfort and minimizing complications.

The ASTS (for Active Scoliosis Treatment System) growing rod is a new fully implantable motorized spinal distraction device which can ensure a correction of scoliosis and progressive elongation ensuring patient comfort and minimizing complications.

DETAILED DESCRIPTION:
Despite a better understanding and technical progress, the evolutionary early scoliosis remains a therapeutic challenge. The definition includes idiopathic scoliosis beginning before the age of 3 years, congenital scoliosis, neuromuscular and syndromic. Spinal deformity is often progressive and may compromise cardiorespiratory function.

The goal of treatment is to prevent further avoiding spinal fusion in a subject in growth. Surgery is indicated in case of failure or cons-indication of conservative treatment (corset or plaster). The principle is to position the posterior rods subcutaneous or in muscle attached to two ends of the deformation.

Intraoperative distraction allows correction of the deformity. A new distraction is performed every 6 months until skeletal maturity.

Considerable complication rates are reported (58%), mainly implant infections and disassembly, because of the need for multiple reoperations. Motorized implants can potentially avoid repeated interventions limiting complications.

Thus, the central hypothesis of this project is a new fully implantable motorized spinal distraction device may provide a correction of scoliosis and progressive elongation ensuring patient comfort and minimizing complications.

ELIGIBILITY:
Inclusion Criteria:

* Patient 4 to 10 years
* Patient weight between 15kg at 50kg
* Introducing severe scoliosis (Cobb angle> 40 °) with early onset
* Failed or cons-indication of conservative treatment (cast or brace)
* Agreement of parents or legal guardian (written agreement) and the patient (at least an oral agreement).

Exclusion Criteria:

* Contraindication to surgery
* Age less than 4 years or above 10 years
* Weight less 15kg and above 50 kg

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Ability to Implant the device | Day 0: the day of the implantation
  The surgeon will have to say if the implantation of the device has been done or not
Change of the position of the implant | 1 years after the implantation
  1 year after the implantation of the device, radiographs will be realised to ensure that the implant is still well positioning
Change of the position of the implant | 2 years after the implantation
  2 years after the implantation of the device, radiographs will be realised to ensure that the implant is still weel positioning
Change of the position of the implant | 3 years after the implantation
  3 years after the implantation of the device, radiographs will be realised to ensure that the implant is still weel positioning
Change of the implant's length | 3 months, 6 months, 9 months, 1 year, 2 years and 3 years after the implantation
  The elongation of the implant will be measured in mm on the digital radiography

SECONDARY OUTCOMES:
Post-surgical pain | 3 months, after the implantation
  Self-assessment of pain using a visual analog scale
Post-surgical pain | months after the implantation
  Self-assessment of pain using a visual analog scale
Post-surgical pain | 9 months after the implantation
  Self-assessment of pain using a visual analog scale
Post-surgical pain | 1 year after the implantation
  Self-assessment of pain using a visual analog scale
Survey to evaluate the quality of life | Day 0
  Assess quality of life in the questionnaire PedsQL
Survey to evaluate the quality of life | 6 months after the implantation
  Assess quality of life in the questionnaire PedsQL
Survey to evaluate the quality of life | 1 year after the implantation
  Assess quality of life in the questionnaire PedsQL
to ease for the surgeon to implant the device, | Day 0
  Number of participant with ease for the surgeon to implant the device,
wound closure without tension, | Day 0
  Number of participant with closure of the wound without tension,
good positioning of the radiographic implant. | Day 0
  Number participant with good positioning of the radiographic implant.
Number of medical visits | 1 year
  Measure of the number of medical visit in the year after implant
Determine the number of iterative extensions made during follow-up | 1 year
  Number of iterative extensions of 1 year.
correction of deformation immediately after the operation, | 3 months, 6 months, 9 month and 1 year
  Number of participant with correction of deformation immediately after the operation,
correction of deformation immediately after the operation, | 3 months after implantation
  Number of participant with correction of deformation immediately after the operation,
Loss correction at 1 year | 6 months after implantation
  Loss correction at 1 year
Loss correction at 1 year | 9 month after implantation
  Loss correction at 1 year
Loss correction at 1 year | 1 year after implantation
  Loss correction at 1 year
Increase the distance T1-S1 at 1 year | 1 year
  Increase the distance T1-S1 at 1 year (in mm)
Effective Elongation measured on radiographs of specification of the device (in mm) | 3 months after implantation
  Effective Elongation measured on radiographs of specification of the device (in mm)
Effective Elongation measured on radiographs of specification of the device | 6 months after implantation
  Effective Elongation measured on radiographs of specification of the device (in mm)
Effective Elongation measured on radiographs of specification of the device | 9 month after implantation
  Effective Elongation measured on radiographs of specification of the device (in mm)
Effective Elongation measured on radiographs of specification of the device | 1 year after implantation
  Effective Elongation measured on radiographs of specification of the device (in mm)
Nature of complications | 1 years
  describe the nature of complication
Nature of complications | 2 years
  describe the nature of complication
Nature of complications | 3 years
  describe the nature of complication
Nature of complications | 5 years
  describe the nature of complication

CONTACTS AND LOCATIONS:
Overall Officials: Franck Accadbled, MD PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU de Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Noordeen HM, Shah SA, Elsebaie HB, Garrido E, Farooq N, Al-Mukhtar M. In vivo distraction force and length measurements of growing rods: which factors influence the ability to lengthen? Spine (Phila Pa 1976). 2011 Dec 15;36(26):2299-303. doi: 10.1097/BRS.0b013e31821b8e16. PMID 21494191
- [Background] Varni JW, Seid M, Kurtin PS. PedsQL 4.0: reliability and validity of the Pediatric Quality of Life Inventory version 4.0 generic core scales in healthy and patient populations. Med Care. 2001 Aug;39(8):800-12. doi: 10.1097/00005650-200108000-00006. PMID 11468499
- [Background] Varni JW, Burwinkle TM, Seid M, Skarr D. The PedsQL 4.0 as a pediatric population health measure: feasibility, reliability, and validity. Ambul Pediatr. 2003 Nov-Dec;3(6):329-41. doi: 10.1367/1539-4409(2003)0032.0.co;2. PMID 14616041
- [Background] Akbarnia BA, Marks DS, Boachie-Adjei O, Thompson AG, Asher MA. Dual growing rod technique for the treatment of progressive early-onset scoliosis: a multicenter study. Spine (Phila Pa 1976). 2005 Sep 1;30(17 Suppl):S46-57. doi: 10.1097/01.brs.0000175190.08134.73. PMID 16138066
- [Background] Bess S, Akbarnia BA, Thompson GH, Sponseller PD, Shah SA, El Sebaie H, Boachie-Adjei O, Karlin LI, Canale S, Poe-Kochert C, Skaggs DL. Complications of growing-rod treatment for early-onset scoliosis: analysis of one hundred and forty patients. J Bone Joint Surg Am. 2010 Nov 3;92(15):2533-43. doi: 10.2106/JBJS.I.01471. Epub 2010 Oct 1. PMID 20889912
- [Background] Lucas G, Bollini G, Jouve JL, de Gauzy JS, Accadbled F, Lascombes P, Journeau P, Karger C, Mallet JF, Neagoe P, Cottalorda J, De Billy B, Langlais J, Herbaux B, Fron D, Violas P. Complications in pediatric spine surgery using the vertical expandable prosthetic titanium rib: the French experience. Spine (Phila Pa 1976). 2013 Dec 1;38(25):E1589-99. doi: 10.1097/BRS.0000000000000014. PMID 24048087
- [Background] Krieg AH, Speth BM, Foster BK. Leg lengthening with a motorized nail in adolescents : an alternative to external fixators? Clin Orthop Relat Res. 2008 Jan;466(1):189-97. doi: 10.1007/s11999-007-0040-3. Epub 2008 Jan 3. PMID 18196392
- [Background] Baumgart R. The reverse planning method for lengthening of the lower limb using a straight intramedullary nail with or without deformity correction. A new method. Oper Orthop Traumatol. 2009 Jun;21(2):221-33. doi: 10.1007/s00064-009-1709-4. PMID 19685230
- [Background] den Uil CA, Bezemer R, Miranda DR, Ince C, Lagrand WK, Hartman M, Bogers AJ, Spronk PE, Simoons ML. Intra-operative assessment of human pulmonary alveoli in vivo using Sidestream Dark Field imaging: a feasibility study. Med Sci Monit. 2009 Oct;15(10):MT137-141. PMID 19789519
- [Background] Kanter KR, Haggerty CM, Restrepo M, de Zelicourt DA, Rossignac J, Parks WJ, Yoganathan AP. Preliminary clinical experience with a bifurcated Y-graft Fontan procedure--a feasibility study. J Thorac Cardiovasc Surg. 2012 Aug;144(2):383-9. doi: 10.1016/j.jtcvs.2012.05.015. Epub 2012 Jun 13. PMID 22698555
- [Background] Kerimaa P, Ojala R, Sinikumpu JJ, Hyvonen P, Korhonen J, Markkanen P, Tervonen O, Sequeiros RB. MRI-guided percutaneous retrograde drilling of osteochondritis dissecans of the talus: a feasibility study. Eur Radiol. 2014 Jul;24(7):1572-6. doi: 10.1007/s00330-014-3161-6. Epub 2014 Apr 17. PMID 24740345
- [Background] Flynn JM, Emans JB, Smith JT, Betz RR, Deeney VF, Patel NM, Campbell RM. VEPTR to treat nonsyndromic congenital scoliosis: a multicenter, mid-term follow-up study. J Pediatr Orthop. 2013 Oct-Nov;33(7):679-84. doi: 10.1097/BPO.0b013e31829d55a2. PMID 23812154